CLINICAL TRIAL: NCT06073184
Title: Weight-loss Drug for Fertility-Sparing Treatment of Atypical Hyperplasia and Grade 1 Cancer of the Endometrium (WE-FiERCE)
Brief Title: Weight-loss Drug for Fertility-Sparing Treatment of Atypical Hyperplasia and Low-grade Cancer of the Endometrium
Acronym: WE-FiERCE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-5042
Record Dates: First submitted 2023-09-12; First posted 2023-10-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Endometrial Cancer; Atypical Hyperplasia
Keywords: Tirzepatide; pIUD
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Tirzepatide; Levonorgestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tirzepatide and Progestin Intrauterine Device (Experimental): All patients will receive a progestin intrauterine device and tirzepatide subcutaneous injections
  Interventions: Drug: Mounjaro; Drug: Mirena

INTERVENTIONS:
Drug: Mounjaro — Weekly subcutaneous injection of 2.5mg tirzepatide at baseline with dose escalation by 2.5mg every 4 weeks to reach 15mg or the maximum tolerated dose, by Week 20
  Other Names: Tirzepatide
Drug: Mirena — Levonorgestrel-releasing Intrauterine System (52mg) to deliver up to 20 mcg levonorgestrel per day
  Other Names: Progestin-releasing intra-uterine device (pIUD)

SUMMARY:
The incidence of endometrial cancer is increasing at an alarming rate. This trend parallels the rising rate of obesity, the most significant risk factor for endometrial cancer. Young women with obesity and endometrial cancer or atypical hyperplasia who want to maintain their fertility are treated with progestin therapy, such as progestin intra-uterine device (pIUD), which is associated with a mediocre response rate and high recurrence rate, and does not address the underlying cause, obesity. Therefore, the investigators want to assess whether the addition of a weight-loss drug to pIUD will improve their oncologic, reproductive and metabolic outcomes.

DETAILED DESCRIPTION:
The research aims to answer the question: "Does the addition of a Glucose-dependent Insulinotropic Polypeptide (GIP)/Glucagon-like Peptide-1 (GLP-1) co-agonist to standard progestin treatment lead to a higher complete response rate compared to historical response rates using progestin alone in young patients with endometrial cancer/atypical hyperplasia who wish to preserve their fertility?".

This is a multicentre single arm open-label phase II clinical trial to assess the complete pathologic response as determined by endometrial sampling after 48 weeks of tirzepatide (GIP/GLP-1 co-agonist) and progestin therapy in patients with BMI ≥ 27 who have endometrial cancer/atypical hyperplasia and desire fertility preservation.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 27
* Diagnosis of grade 1 or 2 endometrioid endometrial cancer or atypical hyperplasia made by either endometrial biopsy or dilation and curettage
* For those with endometrial cancer, clinical FIGO 2009 stage 1A disease without evidence of metastatic disease beyond the uterus and no myometrial invasion by MRI or CT
* ECOG status <2
* Desire for fertility preservation
* Ability to understand and willing to sign a written informed consent document

Exclusion Criteria:

* Evidence of myometrial invasion or extra-uterine disease on imaging
* High grade or p53 mutated (p53mut) endometrial cancer
* Estrogen receptor negative endometrial cancer (positivity defined as moderate/strong staining>10%)
* Mismatch repair deficient (MMRd) endometrial cancer
* History of other malignancies except if curatively treated with no evidence of disease for >5 years
* Previous surgical treatment of obesity
* Current use of weight loss medication (no use in last 2 months)
* Medical co-morbidity with end-organ dysfunction
* Contraindications to pIUD or tirzepatide.
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures.

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 71 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2032-02 (Estimated)

PRIMARY OUTCOMES:
Assessment of Complete Pathologic Response | 48 weeks
  Proportion of patients (%) who achieve pathological complete response at 48 weeks after initiation of pIUD and tirzepatide.

SECONDARY OUTCOMES:
Assessment of Safety and Tolerability | 48 weeks
  Adverse events during treatment period
Assessment of Feasibility | 2.5 years
  Rate of accrual; Patient compliance; Retention
Assessment of Secondary Oncologic Outcomes | 6 years
  Time to achieve complete response; Duration of response; Recurrence rate; Time to recurrence; Progression/persistence rate
Assessment of Reproductive Outcomes | 6 years
  Rate of pregnancy; Live birth; Miscarriage; Pregnancy complications
Assessment of Patient Reported Outcomes | 48 weeks
  Quality of Life; Psychological functioning and fertility concerns after cancer diagnosis
Assessment of Metabolic Outcomes | 48 weeks
  Weight; BMI; Waist/hip circumference; Serum biomarkers of obesity and insulin resistance

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Soyoun Kim, MD, Principal Investigator — University Health Network, Toronto; Sarah E Ferguson, MD, Principal Investigator — University Health Network, Toronto